CLINICAL TRIAL: NCT03587727
Title: Hepatic Fat Content and Mitochondrial Flux in Obese Youth Before and After Bariatric Surgery
Brief Title: Hepatic Mitochondrial Function in Youth
Acronym: MANGO
Status: Completed | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Other Study IDs: 18-0479
Record Dates: First submitted 2018-06-14; First posted 2018-07-16 (Actual); Results first posted 2025-10-10 (Actual); Last update posted 2025-10-10 (Actual); Status verified 2025-09

CONDITIONS: Hepatic Steatosis; Bariatric Surgery Candidate; Adolescent Obesity; Obesity
Keywords: bariatric surgery; hepatic mitochondria; insulin secretion
MeSH Terms: conditions — Fatty Liver; Pediatric Obesity; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — With participant consent, samples will be kept and may be used in future research to learn more about NAFLD and risk for type 2 diabetes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Assess the impact of bariatric surgery on hepatic energy metabolism and glucose and insulin dynamics in obese youth

DETAILED DESCRIPTION:
A metabolic study that will be performed prior to and 12 months following bariatric surgery. The study will include 31-phosphorus magnetic resonance spectroscopy to measure phosphate concentrations in the liver; a 4 hour mixed meal tolerance test, an intravenous arginine test, Abdominal Magnetic Resonance Imaging (MRI) for visceral and hepatic fat, Magnetic Resonance (MR) Elastography of the liver, indirect calorimetry, body composition assessment with Bodpod, serum metabolomics and hepatic tissue mitochondrial measures from the time of surgery only.

ELIGIBILITY:
Inclusion Criteria:

1. Obese youth ages 13-20 years, scheduled for bariatric surgery at Children's Hospital Colorado
2. BMI 35-55 m2/kg
3. Maximal body circumference <200 cm

Exclusion Criteria:

1. Use of medications known to affect insulin sensitivity: oral glucocorticoids within 10; days, atypical antipsychotics, immunosuppressant agents, HIV medications.
2. Infectious hepatitis
3. Alcohol abuse
4. Mitochondrial disease
5. Type 2 diabetes
6. Medications that affect hepatic outcomes (e.g. PPAR-γ or PPAR-α, metformin)
7. Currently pregnant or breastfeeding women. Development of pregnancy during the study period will necessitate withdrawal from the study.
8. Severe illness requiring hospitalization within 60 days
9. Diabetes, defined as Hemoglobin A1C > 6.4%
10. Anemia, defined as Hemoglobin < 10 mg/dL
11. Diagnosed major psychiatric or developmental disorder limiting informed consent
12. Implanted metal devices that are not compatible with MRI

Ages: 13 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Individuals age 13-20 years; Body Mass Index 35-55 m2/kg; Scheduled for Bariatric Surgery at Children's Hospital Colorado.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2018-11-20 (Actual); Primary Completion 2023-06-21 (Actual); Study Completion 2023-06-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Melanie Cree-Green, MD, PhD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Anshutz Medical Campus/Children's Hospital Colorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Teenagers 13-20 Years Old in Bariatric Surgery Program: 13-20 year old male and female participants before and after bariatric surgery.
Period: Overall Study
Arm/Group | Teenagers 13-20 Years Old in Bariatric Surgery Program
Started | 20
Completed | 6
Not Completed | 14
Not completed — 10 did not complete either of the pre-op MMTT or post-op MMTT. | 10
Not completed — 4 completed the pre-op MMTT but did not complete the post-op MMTT. | 4

BASELINE CHARACTERISTICS:
Arm/Group | Teenagers 13-20 Years Old in Bariatric Surgery Program
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 16.85 (1.576)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12
  Not Hispanic or Latino | 8
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 14
  More than one race | 1
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Change in Percentage of Liver Fat Per MRI
Description: Percentage of liver fat at 1 year post-bariatric surgery minus percentage of liver fat prior to bariatric surgery. Liver fat measured with MRI and calculated via the Dixon method as the proton density hepatic fat. A negative value means a decrease in liver fat after bariatric surgery.
Time Frame: Prior to bariatric surgery and 1 year post-bariatric surgery
Measure: Mean (Standard Deviation); unit: percentage of liver fat
Arm/Group | Teenagers 13-20 Years Old in Bariatric Surgery Program
Number analyzed (Participants) | 6
percentage of liver fat | -13.93 (12.89)

2. Primary Outcome: Change in %Direct TG-Glycerol Appearance
Description: Change in %TG-Glycerol appearance from a labeled glycerol drink via direct pathway. TCA substrate cycling assessed via change in fractional direct glycerol carbon contributions to newly synthesized triglycerides using a U-13C glycerol tracer drink. A higher direct percentage is beneficial, indicating decreased oxidative stress resulting from excess glycerol metabolism through the TCA cycle.
Time Frame: Prior to bariatric surgery and 1 year post-bariatric surgery
Measure: Mean (Standard Deviation); unit: change in percentage of Direct TG-Glycer
Arm/Group | Teenagers 13-20 Years Old in Bariatric Surgery Program
Number analyzed (Participants) | 6
change in percentage of Direct TG-Glycer | 0.33 (3.204)

3. Secondary Outcome: Change in Insulin Sensitivity
Description: Mixed meal tolerance test (MMTT): measured with SI. This is a measure of post-prandial (MMTT) insulin sensitivity as calculated with the Oral Minimal Model (OMM) using SAAM II Software. This software uses participant weight, glucose and insulin concentrations at various time points during the MMTT to calculate the participant insulin sensitivity. A positive Si value means an increase in insulin sensitivity.
Time Frame: Prior to bariatric surgery and 1 year post-bariatric surgery
Measure: Mean (Standard Deviation); unit: dL/kg/min/μU/mL
Arm/Group | Teenagers 13-20 Years Old in Bariatric Surgery Program
Number analyzed (Participants) | 6
dL/kg/min/μU/mL | 0.000552758 (0.000634641)

4. Secondary Outcome: Change in Peak Glucose
Description: Mixed meal tolerance test (MMTT): Peak glucose concentration (mg/dL) during 4 hour MMTT with 16 time points.
Time Frame: Prior to bariatric surgery and 1 year post-bariatric surgery
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Teenagers 13-20 Years Old in Bariatric Surgery Program
Number analyzed (Participants) | 6
mg/dL | 11.5 (14.802)

5. Secondary Outcome: Change in Minimum Glucose
Description: Mixed meal tolerance test (MMTT): Minimum glucose concentration (mg/dL) during 4 hour MMTT with 16 time points.
Time Frame: Prior to bariatric surgery and 1 year post-bariatric surgery
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Teenagers 13-20 Years Old in Bariatric Surgery Program
Number analyzed (Participants) | 6
mg/dL | -7 (15.192)

6. Secondary Outcome: Change in Peak Insulin
Description: Mixed meal tolerance test (MMTT): Peak insulin concentration (uIU/mL) during 4 hour MMTT with 13 time points.
Time Frame: Prior to bariatric surgery and 1 year post-bariatric surgery
Measure: Mean (Standard Deviation); unit: uIU/mL
Arm/Group | Teenagers 13-20 Years Old in Bariatric Surgery Program
Number analyzed (Participants) | 6
uIU/mL | 28.333 (62.746)

7. Secondary Outcome: Change in Minimum Insulin
Description: Mixed meal tolerance test (MMTT): Minimum insulin concentration (uIU/mL) during 4 hour MMTT with 13 time points.
Time Frame: Prior to bariatric surgery and 1 year post-bariatric surgery
Measure: Mean (Standard Deviation); unit: uIU/mL
Arm/Group | Teenagers 13-20 Years Old in Bariatric Surgery Program
Number analyzed (Participants) | 6
uIU/mL | -7.333 (3.7771)

8. Secondary Outcome: Change in Peak C-peptide
Description: Mixed meal tolerance test (MMTT): Peak c-peptide concentration (ng/mL) during 4 hour MMTT with 10 time points.
Time Frame: Prior to bariatric surgery and 1 year post-bariatric surgery
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Teenagers 13-20 Years Old in Bariatric Surgery Program
Number analyzed (Participants) | 6
ng/mL | 1.7 (3.2323)

9. Secondary Outcome: Change in Peak GLP-1
Description: Mixed meal tolerance test (MMTT): Peak GLP-1 concentration (pmol/L) during 4 hour MMTT with 9 time points.
Time Frame: Prior to bariatric surgery and 1 year post-bariatric surgery
Measure: Mean (Standard Deviation); unit: pmol/L
Arm/Group | Teenagers 13-20 Years Old in Bariatric Surgery Program
Number analyzed (Participants) | 6
pmol/L | -7.1117 (36.883)

10. Secondary Outcome: Change in Fasting Glucagon
Description: Mixed meal tolerance test (MMT): Fasting glucagon concentration (pg/mL) at the beginning of a 4 hour MMTT 1 year post bariatric surgery minus prior to surgery. A negative value means there was a decrease in fasting glucagon concentrations one year post-bariatric surgery.
Time Frame: Prior to bariatric surgery and 1 year post-bariatric surgery
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Teenagers 13-20 Years Old in Bariatric Surgery Program
Number analyzed (Participants) | 6
pg/mL | -41.333 (32.672)

11. Secondary Outcome: Change in Liver Stiffness Per MRI
Description: Change from baseline in degree of hepatic stiffness, measured with Magnetic Resonance elastography (MRE).
Time Frame: Prior to bariatric surgery and 1 year post-bariatric surgery
Population: Participants that completed pre-op and post-op study visits including valid MRE at each visit.
Measure: Mean (Standard Deviation); unit: kPa
Arm/Group | Teenagers 13-20 Years Old in Bariatric Surgery Program
Number analyzed (Participants) | 4
kPa | -0.234 (0.508)

12. Secondary Outcome: Mitochondrial Function in the Liver Assessed by Oroboros
Description: L/E Coupling Control Ratio: Maximal respiratory capacity was examined in permeabilized hepatic tissue from adolescents using pyruvate (carbohydrate) and palmitoylcarnitine (lipid) as a substrate. Respiratory capacity was normalized to hepatic tissue wet weight. Coupling control ratio (L/E) was calculated as oxygen flux in leak (oligomyocin) divided by ET capacity (FCCP) with a maximum coupling of 1.0.
Time Frame: At the time of surgery
Population: 14 participants completed in-surgery study measures, regardless of participation in pre-op or post-op MMTTs.
Measure: Mean (Standard Deviation); unit: Coupling Control Ratio (unitless)
Arm/Group | Teenagers 13-20 Years Old in Bariatric Surgery Program
Number analyzed (Participants) | 14
Coupling Control Ratio (unitless)
  Carbohydrate L/E Coupling Control Ratio | 0.34 (0.06)
  Lipid L/E Coupling Control Ratio | 0.50 (0.9)

13. Secondary Outcome: Hepatic Steatosis Score Via Tissue Biopsy
Description: NAFLD (non-alcoholic fatty liver disease) Activity Score (NAS) determined via liver tissue biopsy and graded by a pathologist. The NAS can range from 0 to 8 and is calculated by the sum of scores of steatosis (0-3), lobular inflammation (0-3) and hepatocyte ballooning (0-2). A higher number represent a worse outcome.
Time Frame: At the time of surgery
Population: Number of patients that had a liver tissue biopsy.
Measure: Number; unit: participants
Arm/Group | Teenagers 13-20 Years Old in Bariatric Surgery Program
Number analyzed (Participants) | 15
participants
  NAFLD Activity Score: 0 NAS ≤ 3 correlated with a diagnosis of "not NASH" | 3
  NAFLD Activity Score: 1 NAS ≤ 3 correlated with a diagnosis of "not NASH" | 1
  NAFLD Activity Score: 2 NAS ≤ 3 correlated with a diagnosis of "not NASH" | 3
  NAFLD Activity Score: 3 NAS ≤ 3 correlated with a diagnosis of "not NASH" | 4
  NAFLD Activity Score: 4 | 3
  NAFLD Activity Score: 5 NAS score of ≥ 5 strongly correlated with a diagnosis of "definite NASH" | 1

ADVERSE EVENTS:
Time Frame: Duration of study participation, about 1 year.
Arm/Group | Teenagers 13-20 Years Old in Bariatric Surgery Program
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

LIMITATIONS AND CAVEATS:
Limited by small sample size due to participant withdraw.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-02-14): https://cdn.clinicaltrials.gov/large-docs/27/NCT03587727/Prot_SAP_000.pdf